CLINICAL TRIAL: NCT06598527
Title: Stereotactic Body Radiotherapy Followed by Tislelizumab Plus Platinum-based Chemotherapy Versus Tislelizumab Plus Platinum-based Chemotherapy as Neoadjuvant Therapy in Patients With Resectable Stage Ⅱ-Ⅲ Non-small Cell Lung Cancer: A Phase Ⅲ, Randomized, Multicenter, Prospective Study
Acronym: SACTION2401
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yang Hong (Other)
Responsible Party: Sponsor-Investigator, Yang Hong, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-495-01
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer (NSCLC)
Keywords: NSCLC; SBRT; immunochemotherapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; tislelizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- neoadjuvant SBRT combined with immunochemotherapy (Experimental): Following admission, intrapulmonary primary stereotactic body radiotherapy (SBRT) was administered at a dosage of 24 Gy across three fractions. Subsequently, within seven days of completing SBRT, two cycles of Tislelizumab in combination with a platinum-based double-agent chemotherapy regimen were initiated. These cycles were repeated every three weeks. Surgical intervention was scheduled to occur 4-6 weeks (±7 days) after the completion of the second chemotherapy cycle
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT); Drug: Tislelizumab; Drug: Chemotherapy
- neoadjuvant immunochemotherapy (Active Comparator): Three cycles of Tislelizumab in conjunction with platinum-based chemotherapy were administered at three-week intervals. Surgical intervention was subsequently scheduled to occur within 4 to 6 weeks (±7 days) following the completion of the third chemotherapy cycle.
  Interventions: Drug: Tislelizumab; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — Radiation source: 6MV photon linear gas pedal is used. Position immobilization: supine position, hands up, vacuum bag or styrofoam immobilization.
  Radiotherapy plan design: 4DCT positioning, radiotherapy plan design at 20% respiratory time-phase CT, isocentric irradiation, IMRT or VMAT design.
  Definition of target area:
  Gross tumor volume (GTV) includes the primary tumor in the lung, excluding lymph nodes. Internal target volume (ITV); Internal target volume (ITV) is formed by the fusion of 10 respiratory phases of GTV; Planning target volume (PTV) is formed by expanding the ITV by 0.5 cm in all directions.
  Other Names: SBRT
  Arms: neoadjuvant SBRT combined with immunochemotherapy
Drug: Tislelizumab — PD-L1 inhibitor
Drug: Chemotherapy — platinum-based double-agent chemotherapy

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of neoadjuvant Stereotactic Body Radiotherapy (SBRT) combined with immunochemotherapy versus neoadjuvant immunochemotherapy. The main questions it aims to answer are:

Dose SBRT combined with immunochemotherapy improve event-free survival? Is SBRT combined with immunochemotherapy safe enough?

Participants will:

Receive neoadjuvant SBRT combined with immunochemotherapy or neoadjuvant immunochemotherapy.

Tumor assessment will be performed prior to surgery. Surgery will be performed within 4 to 6 weeks (+ 7 days) after completion of the last cycle of immunochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients voluntarily agree to participate and sign the informed consent; 2. Patients with cytologically/histologically diagnosed (by means of percutaneous lung aspiration biopsy, bronchoscopy, mediastinoscopy, etc.), untreated stage IIa-IIIa (according to the AJCC 8th edition of thoracic tumor staging) non-small cell lung cancer. In addition, patients with potentially resectable stage IIIb (T3-4N2) NSCLC will also be enrolled. All patients are required to receive PET/CT (or chest + upper abdominal CT + brain MRI) at baseline for clinical staging; 3. Pulmonary lesions will be assessed as resectable/potentially resectable by a multiple disciplinary team including thoracic surgeon; 4. Eastern Cooperative Oncology Group Performance Status 0 to 1 5. Requirements for hematology: i, neutrophils ≥ 1500 x 109/L; ii, platelets ≥ 100 x 109/L; iii, hemoglobin > 9.0 g/dL; iv, serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min; v, aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 3 x ULN; vi, total bilirubin ≤ 1.5 x ULN; vii. forced expiratory volume in the first second (FEV1) ≥ 1.2 L or > 40% predicted; viii. International Normalized Ratio/activated partial thromboplastin time (INR/APTT) within the normal range; 6. Age 18-75

Exclusion Criteria:

* 1. Patients with or suspected with autoimmune diseases. Note: patients with vitiligo, type 1 diabetes, hypothyroidism managed with hormone replacement therapy only (Hashimoto's thyroiditis) can be enrolled in the study when there is no clear evidence of recurrence; 2. Patients required systemic corticosteroids treatment (dose > 10 mg daily prednisolone [or equivalent]) or other immunosuppressive drugs within 14 days of enrollment. Note: inhaled or topical corticosteroids, or adrenal replacement therapy (dose > 10 mg daily prednisolone [or equivalent]) are acceptable for patients without apparent autoimmune disease; 3. Historical radiotherapy of chest 4. Active bleeding before treatment 5. Patents with sever heart, lung, liver, or kidney insufficiency 6. Diabetes more than 10-year; unsatisfactory blood glucose control 7. Patients with interstitial lung disease or non-infectious pneumonia 8. EGFR-mutations and ALK-fusion positive NSCLC 9. Patients with other prior malignancies (except skin malignancies other than non-melanoma, and carcinoma in situ at the following sites [bladder, stomach, colorectal, endometrium, cervix, melanoma, or breast]) are not eligible for enrollment in this study. However, if the prior malignancies remain in complete response (CR) for ≥ 2 years and no additional anti-cancer therapy is required during the study, such patients are permitted to be enrolled; 10. The patient is medically, psychologically, or physiologically unable to complete the study or to understand the Patient Information Sheet, in the opinion of the investigator; 11. Received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA any other drugs specifically targeting T-cell co-stimulation or immunoregulation pathways; 12. Present active hepatitis B or hepatitis C 13. Patients with positive HIV test results or diagnosed with acquired immunodeficiency disease (AIDS); 14. Hypersensitivity to the investigational product; 15. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
event-free survival | 5 years
  include 2/3/5 event-free survival time

SECONDARY OUTCOMES:
major pathologic response (MPR) rate | 1-year
pathological complete response (PCR) rates | 1-year
R0-resection rate | 1-year
overall survival | 5 years
  2/3/5 years overall survival rate
safety | 1-year
  adverse events rate, postoperative complication rate, mortality rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No